CLINICAL TRIAL: NCT05425420
Title: Pharmacokinetics, Pharmacodynamics, and Safety of a Single Dose Intravenous Methadone in Healthy Adult Volunteers (MTH02)
Brief Title: Single Dose IV Methadone for Post-Op Pain
Acronym: MTH02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kanecia Obie Zimmerman (Other)
Responsible Party: Sponsor-Investigator, Kanecia Obie Zimmerman, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00113821; Pro00106216 (Other: Duke site IRB#)
Record Dates: First submitted 2022-04-15; First posted 2022-06-21 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone

STUDY DESIGN:
Intervention Model Description: Subjects will be studied on one occasion in the Early Phase Research Unit at Duke University Medical Center for administration of drug, collection of blood samples, and measurements of drug effect. Study drug is intravenous methadone hydrochloride Plasma samples collections are obtained up to 96 hr after dosing. Dark-adapted pupil diameter is measured by infrared camera. Responses to thermal skin stimulation are recorded. Respiratory rate and end-tidal carbon dioxide concentrations are measured. Subject self-assessment of methadone effect is performed using verbal analog scales. Blood samples obtained during the study will be analyzed for plasma concentrations of methadone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm, Open label Methadone IV (Experimental): All participants will be treated with Methadone Hydrochloride IV (over 10 minutes) and monitored overnight.
  Interventions: Drug: methadone hydrochloride 0.1mg/kg

INTERVENTIONS:
Drug: methadone hydrochloride 0.1mg/kg — Single dose of methadone hydrochloride administered via intravenous (IV)

SUMMARY:
Single-center, open label, single-session study to evaluate methadone pharmacokinetics and pharmacodynamic in adults.

DETAILED DESCRIPTION:
The Adult Methadone study will be conducted at a single site, Duke Early Phase Research Unity (DEPRU), to enroll 24 participants. Participants will be treated/monitored overnight with Methadone hydrochloride IV (FDA approved and commercially available), with daily follow-up visits for 1 week total. The study aims to provide information on the disposition and clinical effects of intravenous methadone to update the drug label.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to < 40 years of age at the time of enrollment
2. Provide informed consent

Exclusion Criteria:

1. History of cardiac dysfunction
2. History of or current QTc prolongation, defined as > 470 ms in males and > 480 ms in females
3. Known hypersensitivity to methadone hydrochloride or any other ingredient in the methadone hydrochloride injection
4. Known acute bronchial asthma or hypercarbia (known history of known PaCO2 above 45 mm HG)
5. Receipt of a serotonergic drug or buproprion within 7 days prior to study enrollment
6. Receipt of benzodiazepines, muscle relaxants, or other opioids within 7 days prior to study enrollment
7. Receipt of a moderate or strong CYP2B6 inhibitor or inducer - either prescription or non-prescription medications, herbals,34 or foods known to be metabolized by or affecting CYP2B6 - within 30 days prior to study enrollment

   1. CYP2B6 inhibitors include clopidogrel, prasugrel, thioTEPA, ticlopidine, voriconazole, macrolide antibiotics, azole-antifungal agents, fluconazole, Alstonia boonei, Mangifera indica, and Picralima nitida
   2. CYP2B6 inducers include artemisinin antimalarials, barbiturates, carbamazepine, cyclophosphamide, efavirenz, lopinavir, methimazole, nelfinavir, phenobarbital, phenytoin, primidone, rifampicin/rifampin, ritonavir, abacavir, amprenavir, nevirapine, telaprevir
8. Receipt of zidovudine, desipramine, or other drugs that may increase serum concentration when combined with methadone within 30 days prior to study enrollment
9. Known or suspected gastrointestinal obstruction, including paralytic ileus
10. Significant respiratory depression (respiratory rate less than 8 breaths/min or oxygen saturation (SpO2) <95%)
11. BMI ≥ 33 and BMI ≤ 17
12. Known history of moderate-to-severe liver (Child Class B or C) or kidney disease (serum creatinine > 1.5)
13. Known history of drug or alcohol addiction (prior or present addiction or treatment for addiction)
14. Females who are pregnant or nursing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD, MPH,PhD, Principal Investigator — DUMC, DCRI
Locations (1):
- Duke Early Phase Unit (DEPRU, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Methadone IV: All participants will be treated with Methadone Hydrochloride IV (over 10 minutes) and monitored overnight.
  Methadone hydrochloride 0.1mg/kg: Single dose of methadone hydrochloride administered via intravenous (IV)
Period: Overall Study
Arm/Group | Open Label Methadone IV
Started | 22
Completed | 19
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Failure to Meet Continuation Criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) in Adults - Systemic Clearance (CL)
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
liters/hour | 6.14 (1.42)

2. Primary Outcome: Pharmacokinetics (PK) in Adults - Volume of Distribution
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
liters | 318.95 (42.04)

3. Primary Outcome: Pharmacokinetics (PK) in Adults - Elimination Half-life
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
hours | 39.66 (9.95)

4. Primary Outcome: Pharmacokinetics (PK) in Adults - Plasma AUC0-96
Description: Plasma AUC0-96 is the area under the plasma concentration versus time curve from time zero to 96 hours post-dose.
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
ng*h/mL | 1088.9 (311.9)

5. Primary Outcome: Pharmacokinetics (PK) in Adults - AUC0-inf
Description: AUC0-inf is the area under the curve from time 0 extrapolated to infinite time.
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
ng*h/mL | 1363.3 (515.7)

6. Primary Outcome: Pharmacokinetics (PK) in Adults - Cmax
Description: Cmax: A pharmacokinetic measure used to determine drug dosing. Cmax is the highest concentration of a drug in the blood, cerebrospinal fluid, or target organ after a dose is given.
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
ng/mL | 90.92 (38.14)

7. Primary Outcome: Pharmacokinetics (PK) in Adults - Tmax
Description: Tmax is the time corresponding to maximum concentration post-dose.
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
hours | 0.116 (0.095)

8. Primary Outcome: Pharmacokinetics (PK) in Adults - Cmin
Description: Cmin is the observed minimum concentration post-dose.
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
ng/mL | 4.35 (2.41)

9. Primary Outcome: Pharmacokinetics (PK) in Adults - Elimination Rate Constant
Description: Elimination rate constant (ke)-s a value used in pharmacokinetics to describe the rate at which a drug is removed from the human system.
Time Frame: 96 hours after dosing
Population: Participants with samples collected at 96 hours.
Measure: Mean (Standard Deviation); unit: h^-1
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 20
h^-1 | 0.018 (0.004)

10. Secondary Outcome: Pharmacodynamics (PD) in Adults - Dark-adapted Pupillometry
Description: Dark-adapted pupillometry measured pupil diameter using a goggle-based, camera-like device. A goggle-based system effectively allowed the participant to be in the dark while room lights were on for research staff.
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
mm
  Left pupil | 6.95 (1.30)
  Right pupil | 7.57 (1.29)

11. Secondary Outcome: Pharmacodynamics (PD) in Adults - Thermal Pain Tolerance Threshold
Description: The thermal pain tolerance threshold is the highest tolerated temperature change. Thermal pain tolerance was measured by a 3 cm2 computer-controlled Peltier-type thermal stimulator. The stimulator delivered painful heat stimuli to the volar side of the forearm. The thermode system's baseline temperature was set at 32°C. The computer-controlled thermode system was programmed to gradually increase the stimulus (0.8°C/sec) until participants pressed a stop button, which indicates maximum tolerable temperature was reached and initiated immediate thermode cooling. The maximum tolerable temperature was recorded.
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
degrees Celsius | 46.58 (1.87)

12. Secondary Outcome: Pharmacodynamics (PD) in Adults - Subjective Self-assessment of Methadone Effects - Alertness/Sedation
Description: Subjective self-assessment of methadone effects using a visual analog scale (VAS). The score for alertness/sedation ranges from 0 (almost asleep) to 100 (wide awake).
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
score on a scale | 91.60 (16.33)

13. Secondary Outcome: Pharmacodynamics (PD) in Adults - Subjective Self-assessment of Methadone Effects - Energy Level
Description: Subjective self-assessment of methadone effects using a visual analog scale (VAS). The score for energy level ranges from 0 (no energy) to 100 (full of energy).
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
score on a scale | 89.60 (18.01)

14. Secondary Outcome: Pharmacodynamics (PD) in Adults - Subjective Self-assessment of Methadone Effects - Confusion
Description: Subjective self-assessment of methadone effects using a visual analog scale (VAS). The score for confusion ranges from 0 (clear headed) to 100 (confused).
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
score on a scale | 1.60 (3.36)

15. Secondary Outcome: Pharmacodynamics (PD) in Adults - Subjective Self-assessment of Methadone Effects - Clumsiness
Description: Subjective self-assessment of methadone effects using a visual analog scale (VAS). The score for clumsiness ranges from 0 (well-coordinated) to 100 (extremely clumsy).
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
score on a scale | 2.60 (5.37)

16. Secondary Outcome: Pharmacodynamics (PD) in Adults - Subjective Self-assessment of Methadone Effects - Anxiety
Description: Subjective self-assessment of methadone effects using a visual analog scale (VAS). The score for anxiety ranges from 0 (calm/relaxed) to 100 (extremely nervous).
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
score on a scale | 1.50 (3.52)

17. Secondary Outcome: Pharmacodynamics (PD) in Adults - Subjective Self-assessment of Methadone Effects - Nausea
Description: Subjective self-assessment of methadone effects using a visual analog scale (VAS). The score for nausea ranges from 0 (no nausea) to 100 (worst nausea).
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
score on a scale | 0.0 (0.0)

18. Secondary Outcome: Pharmacodynamics (PD) in Adults - Maximum End-expired CO2 Concentration
Description: Measured in mmHg
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
mmHg | 37.40 (1.91)

19. Secondary Outcome: Pharmacodynamics (PD) in Adults - Maximum Sedation Score
Description: Maximum sedation score obtained via the Modified Observer's Assessment of Alertness/Sedation (MOAA/S). The MOAA/S has a scale of 0 to 5, where 0 = "Does not respond to painful trapezius squeeze" and 5 = "Responds readily to name spoken in normal tone".
Time Frame: 96 hours after dosing
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Methadone IV
Number analyzed (Participants) | 19
score on a scale | 5.0 (0.0)

ADVERSE EVENTS:
Time Frame: Up to 96 hours (4 days)
Arm/Group | Open Label Methadone IV
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 10/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Methadone IV (N=22)
Nausea (Gastrointestinal disorders) | 6
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 1
Blood pressure diastolic abnormal (Investigations) | 1
Blood pressure increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Injection site pain (General disorders) | 1
COVID-19 (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT05425420/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT05425420/ICF_000.pdf